CLINICAL TRIAL: NCT03785132
Title: Relationship Between Performance Measurement of Intraoperative Mean Arterial Pressure and Mortality in Patients Undergoing Cardiac Surgery
Brief Title: Performance Measurement in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Youn Joung Cho, MD, Clinical assistant professor, Seoul National University Hospital
Other Study IDs: PM_cardiac surgery
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Blood Pressure
Keywords: blood pressure; performance measurement; cardiac surgery; mortality
MeSH Terms: interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cardiac surgery: Patients who underwent cardiac surgery with cardiopulmonary bypass
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery — The relationship between performance measurement of blood pressure during cardiac surgery (before, during and after cardiopulmonary bypass) and postoperative mortality

SUMMARY:
This study aimed to evaluate the relationship between the perioperative blood pressure and postoperative mortality after cardiac surgery using performance measurement (PM) of mean arterial pressure (MAP).

DETAILED DESCRIPTION:
The authors conducted a retrospective cohort study of adult patients who underwent cardiac surgery requiring cardiopulmonary bypass (CPB). Median performance error (MDPE), median absolute performance error (MDAPE), and wobble of MAP were calculated using preoperative MAP as the reference value, and MBPs before, during and after the bypass as measured values. Univariable and multivariable logistic regression analyses were performed using PM parameters to predict in-hospital mortality. Survival after cardiac surgery was compared using the Cox proportional hazard model. Predictability of PM was assessed using the area under the receiver-operating characteristic curve (AUROC).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery with cardiopulmonary bypass between 2013 and 2016 at Seoul National University Hospital.

Exclusion Criteria:

* Patients without information on preoperative blood pressure or mortality.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery with cardiopulmonary bypass between 2013 and 2016 at Seoul National University Hospital
Sampling Method: Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Mortality | through study completion, average 3 years
  mortality after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Youn Joung Cho, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lee HC, Ryu HG, Jung CW. Performance measurement of intraoperative systolic arterial pressure to predict in-hospital mortality in adult liver transplantation. Sci Rep. 2017 Aug 1;7(1):7030. doi: 10.1038/s41598-017-07664-0. PMID 28765633
- [Derived] Yoon S, Park JB, Lee J, Lee HC, Bahk JH, Cho YJ. Relationship between blood pressure stability and mortality in cardiac surgery patients: retrospective cohort study. J Clin Monit Comput. 2021 Aug;35(4):931-942. doi: 10.1007/s10877-020-00631-7. Epub 2021 Jan 3. PMID 33389355